CLINICAL TRIAL: NCT02556229
Title: Phase II Study Evaluating the Efficacy of Aflibercept for the Treatment of Inflammatory Choroidal Neovascularization (CNV) in Young Patients.
Brief Title: Study Evaluating the Efficacy of Aflibercept for the Treatment of Inflammatory CNV in Young Patients (ALINEA).
Acronym: ALINEA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL14_0201; 2014-003695-23 (EudraCT Number)
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Choroidal Neovascularization
Keywords: Aflibercept; inflammatory choroidal neovascularization; young patient
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aflibercept (Experimental): Intravitreal injection of aflibercept (EYLEA) / 2mg
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — The patients are followed on a monthly basis until 52 weeks. Intravitreal injections of aflibercept at a dosage of 2 mg are initiated at inclusion (mandatory injection) with reinjection every 4 weeks only in case of CNV activity (PRN regimen) until 52 weeks.Therefore, each patient receives between 1 and 13 injections in the whole study.

SUMMARY:
Inflammatory choroidal neovascularization (InCNV) is the third cause of CNV after myopia and Age-related Macular Degeneration (AMD). InCNV is a rare but severe disease and its treatment should not be delayed.

InCNV is treated at the moment with off-label anti-VEGF (Vascular Endothelial Growth Factor) therapy and could also benefit from aflibercept (EYLEA), a new anti-VEGF currently indicated in AMD. Case reports suggest that such patients would not need as many injections as in AMD.

ALINEA is an open-label, single arm, prospective, multicenter, phase II study. The main objective is to demonstrate the effectiveness in clinical terms after 52 weeks of treatment with aflibercept on the visual acuity of patients affected by InCNV. A specific dosage regimen is designed to achieve maximum efficiency. The patients are followed on a monthly basis until 52 weeks. The first injection is mandatory. The other ones are injected only in case of active InCNV.

ELIGIBILITY:
Inclusion Criteria:

* 18 < Age < 60 years old
* Patient who give voluntary signed informed consent
* Patient affiliated with the French universal health care system or similar
* Patient with inflammatory CNV, whatever the cause, including multifocal choroiditis, punctate inner choroidopathy, ocular toxoplasmosis, serpiginous choroiditis or Birdshot chorioretinopathy with active primary subfoveal, retrofoveal or juxtafoveal lesions that affect the fovea as evidenced by angiography (fluorescein and/or indocyanine green) and/or SD-OCT in the studied eye
* Patient willing, committed and able to return for all clinic visits and complete all study-related procedures

Exclusion Criteria:

* Pregnant women
* Sexually active men or women of childbearing potential who are unwilling to practice adequate contraception during the study
* Patient who is protected adults according to the terms of the law (French public health laws)
* Involvement in another clinical trial (studied eye and/or the other eye)
* Patient with non-inflammatory CNV, especially:

  * AMD
  * drusen associated with neovessel
  * High myopia defined as refraction ≥ - 6 diopters
* Other curative treatment of inflammatory CNV in the studied eye during the last 3 months before the first intravitreal injection: anti-VEGF therapy, juxta- or extra-foveal macular laser, photodynamic therapy, surgery, external radiotherapy, transpupillary thermotherapy ...
* Medical history of retrofoveal focal macular laser photocoagulation in the studied eye
* Subretinal hemorrhage reaching the fovea center or with a size > 50% of the lesion area
* Fibrosis or retrofoveal retinal atrophy in the studied eye
* Retinal pigment epithelial tear reaching the macula in the studied eye
* Medical history of intravitreal medical device in the studied eye
* Medical history of auto-immune or idiopathic uveitis
* Proved diabetic retinopathy
* Intra-ocular pressure ≥ 25 mmHg despite two topical hypotonic treatments
* Aphakia or lack of lens capsule (not removed by YAG (yttrium aluminium garnet) laser) in the studied eye
* Arterial hypertension that is not controlled by an appropriate treatment and defined by one measure of systolic blood pressure > 180mmHG or 2 consecutive measures > 160mmHg, or by a diastolic blood pressure > 100mmHg
* Antecedents of cerebrovascular disease or myocardial infarction during the last 6 months before inclusion (J1)
* Antecedents of any pathology, metabolic disease, or any serious suspicion of disease during the clinical or laboratory exam that would contraindicate the use of the product, could affect the interpretation of the study results or lead to major risks of complication for the subject
* Renal insufficiency requiring dialysis or renal transplantation
* Previous (less than a year) or actual treatment with systemic administration of anti-VEGF therapy
* Known hypersensitivity to aflibercept, or another drug composite of the medicinal product used; allergy to fluorescein, indocyanine green, anaesthetic eye drops
* Active or suspected ocular or peri-ocular infection
* Medical history of intra-ocular surgery within 28 days before the first injection in the studied eye
* Any illness or ocular condition that would require an intra-ocular surgery in the studied eye within 12 months after the inclusion
* Follow up not possible during 12 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Mean change in best-corrected visual acuity (BCVA) expressed as number of letters gained or lost measured with Early Treatment Diabetic Retinopathy Study (ETDRS) scale from baseline to week 52 | 52 weeks
  BCVA is measured on the ETDRS scale at an initial distance of 4 meters

SECONDARY OUTCOMES:
Mean change in BCVA expressed as number of letters gained or lost measured with ETDRS scale from baseline to week 24 | 24 weeks
Percentage of patients with a <15-letter loss in BCVA measured with ETDRS scale from baseline to week 24 | 24 weeks
Percentage of patients with a <15-letter loss in BCVA measured with ETDRS scale from baseline to week 52 | 52 weeks
Number of injections per patient | 52 weeks
Mean time between 2 injections | 52 weeks
Mean change in central retinal thickness (CRT) in micrometers measured with Spectral Domain - Optical Coherence Tomography (SD-OCT) from baseline to week 24 | 24 weeks
Mean change in central retinal thickness (CRT) in micrometers measured with Spectral Domain - Optical Coherence Tomography (SD-OCT) from baseline to week 52 | 52 weeks
Mean change in neovascular lesion size measured with fluorescein and/or indocyanine green angiography from baseline to week 52 | 52 weeks
Side-effects observed during the study | 52 weeks
Mean change in neovascular lesion morphology measured with fluorescein and/or indocyanine green angiography from baseline to week 52 | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon / Hopital de la Croix Rousse, Lyon, France

REFERENCES:
- [Result] Kodjikian L, Abukhashabah A, Fardeau C, Tadayoni R, Brezin A, Dumas S, Weber M, Bernard L, Loria O, Decullier E, Huot L, Mathis T. Efficacy and safety of Aflibercept for the treatment of inflammatory choroidal neovascularization: The ALINEA study. Acta Ophthalmol. 2023 Feb;101(1):e43-e49. doi: 10.1111/aos.15214. Epub 2022 Jul 13. PMID 35822428